CLINICAL TRIAL: NCT01493102
Title: Incidence of Hypotension Based on the Discontinuation Order of Vasopressors in the Management of Septic Shock
Brief Title: Discontinuation Order of Vasopressors in Septic Shock
Acronym: DOVSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility by interim analysis
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kyeongman Jeon, Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2011-09-007
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Septic Shock
Keywords: septic shock; norepinephrine; vasopressin; hypotension
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus; Hypotension | interventions — Vasopressins; Norepinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vasopressin (Active Comparator): Vasopressin will be reduced first (0.01 U/hour)
  Interventions: Drug: Vasopressin
- Norepinephrine (Active Comparator): Norepinephrine: Norepinephrine will be reduced first (0.1 microgram/kg/hour)
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Vasopressin — Vasopressin will be reduced first (0.01 U/hour)
  Arms: Vasopressin
Drug: Norepinephrine — Norepinephrine will be reduced first (0.1 microgram/kg/hour)
  Arms: Norepinephrine

SUMMARY:
The purpose of this study is to evaluate the incidence of hypotension based on the discontinuation order of norepinephrine and vasopressin in patients receiving concomitant norepinephrine and vasopressin infusions for the treatment of septic shock.

DETAILED DESCRIPTION:
There are little data regarding the discontinuation of vasopressors in patients with septic shock. Therefore, the investigators intend to evaluate the incidence of hypotension based on the discontinuation order of norepinephrine and vasopressin in patients receiving concomitant norepinephrine and vasopressin infusions for the treatment of septic shock.

ELIGIBILITY:
Inclusion Criteria:

* patients 20 years of age or older
* patients of receiving concomitant therapy with norepinephrine and vasopressin for teh management of septic shock
* patients began to reduce the vasopressor

Exclusion Criteria:

* patients who expired or had care withdrawn while receiving norepinephrine and vasopressin
* patients being transferred into the ICU from an outside facility or the operating room
* patients who are suspected to have vasopressin deficiency (eg. HPA axis dysfunction, empty sella)
* acute myocardial infarction or Congestive heart failure (NYHA functional classification III or IV)
* acute mesenteric ischemia
* patients who were received other vasopressor except for norepinephrine or vasopressin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | One hour after dose reduction of vasopressors
  Hypotension is defined as mean arterial pressure is less than 65mmHg

SECONDARY OUTCOMES:
Time of hypotension | One hour after dose reduction of vasopressors
  Time interval (min) from time of dose reduction of vasopressors to time to development of hypotension
Vasopressor free day | 28 days after dose reduction of vasopressors
28-day mortality | 28 days
  All cause mortality within 28 days after hospitalization
ICU mortality | 3 months
  All cause mortlity during ICU admission
In-hospital mortality | 3 months
  All cause mortality during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: kyeongman Jeon, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jeon K, Song JU, Chung CR, Yang JH, Suh GY. Incidence of hypotension according to the discontinuation order of vasopressors in the management of septic shock: a prospective randomized trial (DOVSS). Crit Care. 2018 May 21;22(1):131. doi: 10.1186/s13054-018-2034-9. PMID 29784057